CLINICAL TRIAL: NCT00006412
Title: A Prospective, Multicenter, Randomized Trial Comparing the Efficacy and Safety of Fenofibrate Versus Pravastatin in HIV-Infected Subjects With Lipid Abnormalities
Brief Title: Safety and Effectiveness of Fenofibrate and Pravastatin in HIV-Positive Patients With Abnormal Blood Lipids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5087; 10917 (Registry Identifier: DAIDS ES); ACTG A5087; AACTG A5087
Record Dates: First submitted 2000-10-13; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: Hyperlipidemia; Procetofen; Pravastatin; Antilipemic Agents
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Hyperlipidemias | interventions — Pravastatin; Fenofibrate

INTERVENTIONS:
Drug: Pravastatin sodium
Drug: Fenofibrate

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of fenofibrate and pravastatin in treating HIV-positive patients who have abnormal levels of fat (lipids) in the blood.

Increased lipids in the blood associated with HIV infection and anti-HIV drugs is a growing problem. The drugs used in this study are known to reduce certain lipids, but little is known about their safety and effectiveness. This study will see if one of the drugs is safer and more effective than the other, or if combining the drugs is the safest and most effective way to lower lipids. This study has been changed. On June 26, 2001, this study was reviewed by the Data and Safety Monitoring Board (DSMB). The DSMB is an independent board monitoring the progress of the study. The review showed that neither pravastatin nor fenofibrate alone were effective in reaching all the cholesterol and triglyceride goals. There were no safety concerns. It is not known if the combination of fenofibrate and pravastatin is effective and safe. Therefore, it is important to continue this study.

DETAILED DESCRIPTION:
Lipid disorders associated with HIV infection and antiretroviral therapy are of growing concern. There is little information available on the safety and efficacy of statins or fibrates in the treatment of HIV-associated hyperlipidemias. Fenofibrate and pravastatin both are able to reduce low-density lipoproteins (LDL) and triglycerides (TG), but it is unclear whether one therapy will be more effective than the other, or if combination therapy will be needed to achieve desirable reductions in both LDL and TG. [AS PER AMENDMENT 12/13/01: The NIAID HIV Therapeutic Trials Data and Safety Monitoring Board (DSMB) met June 26, 2001 to review the interim results. The interim monitoring plan for this study states that accrual into either single-agent therapy arm should stop if the response rate failed to meet a pre-specified minimum at the time of interim review. The DSMB found that this stopping criterion was met for each single-therapy arm. The DSMB recommended that patients currently on single-agent therapy be offered the opportunity to initiate dual-agent therapy, regardless of time on study. There were no safety concerns.]

Patients are randomized to either Arm A or Arm B and stratified by gender, TG level, and number of cardiovascular risk factors. Patients add daily fenofibrate (Arm A) or pravastatin (Arm B) to their antiretroviral therapy for 48 weeks. Evaluations at Week 12 determine LDL, TG, and high-density lipid (HDL) levels. Patients who achieve clinical goals for these levels stay on the drug for the rest of the study. Patients who do not achieve the goals by Week 12 receive a combination of pravastatin and fenofibrate for the rest of the study. At regular clinic visits, patients have physical exams and are questioned about their medications, diet, and exercise. Blood samples are drawn for clinical evaluations, including lipid profiles and HIV-1 RNA monitoring. [AS PER AMENDMENT 12/13/01: On June 26, 2001, the DSMB reviewed interim results and determined that the response rates for both arms met the stopping rule for futility. As a result, all patients who were currently on single-agent therapy were offered the opportunity to initiate dual-agent therapy regardless of time on study. No additional accrual was sought; however, exceptions were made for patients who were in screening at the time of the DSMB review. These patients were given the option of starting single- or dual-agent therapy. The DSMB recommended that all patients on dual-agent therapy be followed for 32 weeks to obtain additional safety and efficacy data. Further endpoints will be analyzed after Week 12 of single-agent therapy or Week 32 of dual-agent therapy.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Are on a lipid-lowering diet based on the patient's statement and have been exercising for at least 30 days before being screened for the study. Patients will be asked if they were counseled by their health care provider. The lipid-lowering diet and exercise program do not have to be prescribed by a physician.
* Have a triglyceride (TG) level of at least 200 mg/dl and low-density lipoprotein (LDL) level of at least 130 mg/dl after fasting for 8 to 12 hours.
* Have been treated with anti-HIV drugs for more than 6 months. Patients must be taking the anti-HIV drugs regularly for at least 4 weeks before they enter the study. Patients must be taking anti-HIV drugs regularly for at least 8 weeks if they have changed from taking protease inhibitor (PI) anti-HIV drugs to non-PI anti-HIV drugs. Any combination without a PI must lower the patient's HIV viral levels, as determined by the patient's physician.
* Are willing, if able to become pregnant, to use 2 reliable types of birth control while taking the study drug(s) and for 1 month after stopping the drug(s).
* Have a negative pregnancy test.
* (This reflects a change in inclusion requirements.)

Exclusion Criteria

Patients will not be eligible for the study if they:

* Have a history of heart disease.
* Have uncontrolled high blood pressure within 4 weeks of study entry.
* Have liver disease.
* Have gall bladder disease or symptoms within 3 months prior to study entry or symptoms of gallstones.
* Had surgery to remove their gallbladder within 3 months prior to study entry.
* Have diabetes requiring drug treatment or diabetes not controlled by diet.
* Have hypothyroidism (low thyroid activity).
* Are allergic or sensitive to the study drug(s) or to other lipid-lowering drugs.
* Have rhabdomyolysis (a muscle disease).
* Have taken any prescription or non-prescription lipid-lowering drug within 14 days prior to study entry or for over 24 weeks in the past.
* Take prescription lipid-lowering agents, other than those given by the study, and non-prescription lipid-lowering agents such as garlic supplements.
* Have failed previous statin or fibrate therapy (after 24 weeks of treatment) or have had side effects from these drugs.
* Receive or have received (within 14 days of study entry) treatment not approved by the FDA. Anti-HIV medications and immune-based treatments not approved by the FDA may be allowed on a case-by-case basis with the approval of the protocol team.
* Were given systemic chemotherapy for cancer other than Kaposi's sarcoma (KS).
* Were given radiation therapy within 30 days of study entry.
* Take drugs that increase risk of muscle disease (such as cyclosporine, erythromycin, itraconazole, and ketoconazole), within 14 days of study entry.
* Take or have taken levothyroxine and liothyronine for hypothyroidism.
* Take high doses of testosterone.
* Take creatine monophosphate or drugs that affect the immune system, within 30 days of study entry.
* Abuse drugs or alcohol, and the doctor thinks this may interfere with the study.
* Are pregnant or breast-feeding.
* Had a scheduled anti-HIV treatment withdrawal prior to study entry.
* (This reflects a change in exclusion requirements.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630
Dates: Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aberg, Study Chair
Locations (58):
- United States (57):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Univ of California San Francisco, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Denver Dept of Health and Hosps, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Tripler Army Med Ctr, Tripler AMC, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Community Health Network Inc, Rochester, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hosp / Brown Univ, Providence, Rhode Island
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Julio Arroyo, West Columbia, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Result] Aberg JA, Zackin RA, Brobst SW, Evans SR, Alston BL, Henry WK, Glesby MJ, Torriani FJ, Yang Y, Owens SI, Fichtenbaum CJ; ACTG 5087 Study Team. A randomized trial of the efficacy and safety of fenofibrate versus pravastatin in HIV-infected subjects with lipid abnormalities: AIDS Clinical Trials Group Study 5087. AIDS Res Hum Retroviruses. 2005 Sep;21(9):757-67. doi: 10.1089/aid.2005.21.757. PMID 16218799
- [Result] Evans SR, Fichtenbaum CJ, Aberg JA; A5087 Study Team. Comparison of direct and indirect measurement of LDL-C in HIV-infected individuals: ACTG 5087. HIV Clin Trials. 2007 Jan-Feb;8(1):45-52. doi: 10.1310/hct0801-45. PMID 17434848
- [Result] Fichtenbaum CJ, Yeh TM, Evans SR, Aberg JA. Treatment with pravastatin and fenofibrate improves atherogenic lipid profiles but not inflammatory markers in ACTG 5087. J Clin Lipidol. 2010 Jul-Aug;4(4):279-87. doi: 10.1016/j.jacl.2010.04.003. PMID 20824151